CLINICAL TRIAL: NCT05761951
Title: Phase 2 Study Evaluating the Efficacy of the Combination of DKN-01 (DKK1 Inhibitor, Leap Therapeutics) and Pembrolizumab in the Treatment of Advanced or Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Leap Therapeutics, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0526; NCI-2023-01855 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DKN-01 (Experimental): Participants will receive DKN-01 by vein over about 30 minutes to 2 hours on Day 1 of each cycle, as well ason Day 15 of Cycle 1.
  Interventions: Drug: DKN-01; Drug: Pembrolizumab
- Pembrolizumab (Experimental): Participants will receive pembrolizumab by vein over about 30 minutes on Day 1 of each cycle for up to 24 months.
  Interventions: Drug: DKN-01; Drug: Pembrolizumab

INTERVENTIONS:
Drug: DKN-01 — Given by IV (vein)
Drug: Pembrolizumab — Given by IV (vein)

SUMMARY:
To learn if the combination of DKN-01 and pembrolizumab can help to control advanced or recurrent endometrial cancer.

DETAILED DESCRIPTION:
Primary Objective:

--The primary objective is to determine the efficacy (objective response rate, ORR) of the combination of DKN-01 and pembrolizumab in the treatment of women with advanced, recurrent endometrioid endometrial cancer or non-endometrioid endometrial cancer with a Wnt/ β-catenin activating mutation.

Secondary Objective:

--Estimate clinical benefit, progression-free survival, overall survival, and duration of response in patients with recurrent or progressive EC treated with DKN-01/ Pembrolizumab. To assess the tolerability of the combination.

Exploratory Objective:

* We will perform the following translational studies to determine the correlation between molecular characteristics and likelihood of response to therapy. The six-month progression free survival (PFS) and the median survival from time of study entry (first treatment) to progression (PFS) or death (OS) will be estimated.
* Determine if DKK1 over-expression, using RNAscope in situ hybridization performed in a central lab, is associated with CTNNB1 mutation or mutation in other genes associated with Wnt/β-catenin pathway activation. High expression of DKK1 is defined as greater than 10% positive cells on RNAscope.
* Determine if mutation status of CTNNB1 or other genes known to result in activation of WNT/β-catenin signaling, such as RNF-43, APC, AXIN1/2, RSPO2/3, and ZNRF3 [1], correlate to response to the combination in women with advanced or recurrent EC. Mutation status of these genes will be determined by next-generation sequencing (Oncomine, ThermoFisher) in a CLIA- and CAP-approved Molecular Diagnostics Laboratory in the Division of Pathology & Laboratory Medicine, MD Anderson Cancer Center using formalin-fixed, paraffin-embedded tissues OR other commercially available, CLIA-certified platforms including but not limited to FoundationOne, Tempus, or CARIS. The presence of a mutation in any of these genes will be considered as indicative of Wnt/β-catenin pathway activation in a patient's tumor. Mutation status will be correlated with treatment response. Mutation status will be correlated with tumoral DKK1 expression. NGS will be performed on baseline biopsies of metastatic disease at the time of enrollment, when available, or using the primary tumor from the hysterectomy if tissue cannot be obtained or is inadequate for testing.
* Determine optimal threshold of DKK1 expression and correlation to treatment response to DKN-01 and pembrolizumab.
* Determine if IHC nuclear localization of mutant β-catenin correlates to treatment response to DKN-01 and pembrolizumab.
* Determine if IHC CD73 expression levels correlate to treatment response to DKN-01 and pembrolizumab.
* Determine if PD-L1 IHC levels correlate to treatment response.
* Determine if additional genetics by NGS including but not limited to PIK3CA mutations and TMB correlate to treatment response
* Determine if blood-based protein markers including but not limited to cytokines at baseline and changes on treatment correlate to response

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Female participants age ≥ 18 years at the time of signing informed consent.
3. Must have histologically confirmed diagnosis of advanced or recurrent endometrioid endometrial cancer that is deemed non-curable with either surgery or radiation therapy. Mixed endometrioid patient will be allowed if the endometrioid component is greater than 50% of the tumor and does not include serous or carcinosarcoma. Non-endometrioid endometrial cancer must have a confirmed Wnt-activating mutation (CTNNB1, RNF-43, APC, AXIN1/2, RSPO2/3, and ZNRF3).
4. Patients may have received up to 2 prior systemic therapies for recurrent disease. Note: Chemotherapy given in conjunction with radiation or as part of primary therapy does not count as prior systemic therapy for recurrence. Hormonal therapy does not count toward prior therapy.
5. Must consent to allow for a pre-treatment tumor biopsy. Tumor material from biopsies done before the screening period are acceptable if the biopsy was performed within 3 months prior to the planned treatment start and no other systemic cancer therapy was administered in the interim. If a biopsy is performed as part of the study and the specimen is considered non-diagnostic or does not have enough tissue (occurs less than 10% of the time), archival tissue can be used to determine the study cohort and the patient can still participate in the trial.
6. Must not have received/progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies.
7. Patients must be off all other anti-tumor therapies (including immunologic agents) for at least four weeks prior to start of treatment. Patients on hormonal agents require a washout for 10 days
8. Patients must be off all other anti-tumor therapies (including immunologic agents) for at least four weeks prior to study registration. Patients on hormonal agents require a washout for 10 days
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
10. Women of childbearing potential (WoCBP) must be permanently or surgically sterilized (undergone a total hysterectomy, bilateral lubal tigation, or bilateral oophorectomy) or are postmenopausal for greater than 12 months. (If uncertain of amenorrhea for 12 months, a pregnancy test will be done to confirm pregnancy status.) If ovaries are present and were not previously menopausal at the time of hysterectomy, should have a serum estradiol <10 pm/mL to confirm ovarian senescence.
11. Adequate hematological organ function laboratory values are defined below:

    * Absolute neutrophil count (ANC) ≥1500/µL
    * Platelets ≥100 000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
12. Adequate renal organ function laboratory values are defined below:

    • Creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) of ≤1.5 × ULN OR

    ≥30 mL/min with creatinine levels >1.5 × institutional ULN
13. Adequate hepatic organ function laboratory values are defined below:

    * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN unless liver metastasis are present, in which case it must be ≤5 × ULN
14. Adequate coagulation function laboratory values of international normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) of ≤1.5 × ULN receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
15. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
16. Creatinine clearance (CrCl) should be calculated per institutional standard. Laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

1. Have uterine sarcomas, carcinosarcomas, serous tumors (any component) or pure clear cell carcinomas without documentation of a Wnt-activating mutation (see Figure 2 for definition)
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Previously treated with an anti-DKK1 therapy.
4. Has deficient mismatch repair (dMMR) or microsatellite instability (MSI-H) are excluded.
5. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to enrollment.
6. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAEv5.0 Grade <1 (Exception to this criterion: any grade of alopecia is eligible for the study).
7. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
8. Major surgical procedures, open biopsy or significant traumatic injury within 4 weeks prior to treatment start (minor procedures within 1 week)
9. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. (Note: Administration of killed vaccines is allowed.)
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are eligible.
13. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging. Note: repeat imaging should be performed during study screening. Participants must be clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Note: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
16. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
17. Has an active infection requiring systemic therapy.
18. Has known history of human immunodeficiency virus (HIV) unless patient meets the following criteria:

    1. HIV RNA is undetected
    2. Have hepatitis B surface antigen
    3. Have hepatitis C antibodies unless hepatitis C virus ribonucleic acid (RNA) is undetected/negative).
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Has had an allogenic tissue/solid organ transplant.
22. Has New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
23. Have Fridericia-corrected QT interval (QTcF) >470 msec, or history of congenital long QT syndrome. Any ECG abnormality that in the opinion of the Investigator would preclude safe participation in the study; patients with pacemakers where QTc is not a reliable measure will require an evaluation by a cardiologist to exclude co-existing cardiac conditions which would prohibit safe participation in the study.
24. History of osteonecrosis of the hip or evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan that are symptomatic and clinically significant. Degenerative changes of the hip joint are not exclusionary. Screening of asymptomatic patients is not required.
25. Clinically-significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis.
26. Women of childbearing potential (WoCBP) or who are pregnant or breastfeeding are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org